CLINICAL TRIAL: NCT02654184
Title: Right Lateral Positioning and Its Effect on Induction of General Anesthesia for Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB000087118
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
Keywords: Right lateral; Induction; Children; Anesthesia
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supine group (Active Comparator): Anesthesia induction with sevoflurane for the patient while he is in supine position.
  Interventions: Procedure: supine position
- Right lateral group (Active Comparator): Anesthesia induction with sevoflurane for the patient while he is in right lateral position position.
  Interventions: Procedure: Right lateral position

INTERVENTIONS:
Procedure: supine position — Anesthesia induction with sevoflurane for the patient while he is in supine position.
  Arms: Supine group
Procedure: Right lateral position — Anesthesia induction with sevoflurane for the patient while he is in right lateral position.
  Arms: Right lateral group

SUMMARY:
The quality of induction with sevoflurane, along with its ability to generate optimal conditions for Laryngeal Mask Airway (LMA) insertion without supplemental opioids or muscle relaxants, has also been well documented. An ideal inhalation induction technique besides being rapid and comfortable for the patient should be economical. To achieve rapidity, use of vital capacity breaths with 8% sevoflurane is a more popular method of induction compared with the conventional incremental induction.

DETAILED DESCRIPTION:
100 pediatric patients (age range, 1 to 8 years) scheduled for lower abdominal surgery under anesthesia will be included. All children in both groups will be premedicated with midazolam, 0.5 mg/kg orally, about 30 minutes before the induction of anesthesia. A parent or guardian accompanied the child into the operating room to allow the child to remain calm and cooperative for inhalation induction. Before induction, pulse oximetry and electrocardiogram monitoring will be attached. For each group, inhalation induction was initiated using a face mask using "tidal volume" and "vital capacity" breathing in high sevoflurane concentration (8%).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 years to 8 years
* Children with ASA class I/II and their willingness to participate in the study

Exclusion Criteria:

* Known seizure disorder
* Craniofacial abnormalities/difficult airway
* Cardiopulmonary or neuromuscular defects
* Hepatic or renal insufficiency
* Expected difficult intravenous (IV) cannulation (eg, dark complexion, obese)
* Catching colds during the past four weeks

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Induction time | an expected 30 minutes
  The time from starting induction of anesthesia until successful insertion of the LMA (seconds)

SECONDARY OUTCOMES:
LMA trials (Number of patients in each group required insertion of an LMA more than once) | an expected 60 minutes
  Number of patients in each group required insertion of an LMA more than once
Blood pressure | Duration of from starting induction of anesthesia till LMA an expected average of 60 minutes
  Systolic, diastolic and mean blood pressure "mm Hg"
Heart rate | Duration of from starting induction of anesthesia till LMA an expected average of 60 minutes
  Heart rate "beats per minute"
Oxygen saturation | Duration of from starting induction of anesthesia till LMA an expected average of 60 minutes
  Oxygen saturation %

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided